CLINICAL TRIAL: NCT06738186
Title: "Bliib Fit - Mach Mit!" in Alters- Und Pflegeinstitutionen
Brief Title: "Bliib Fit - Mach Mit!" in Residential Care Facilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Switzerland University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Eling de Bruin, Prof., Eastern Switzerland University of Applied Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-01990
Record Dates: First submitted 2024-11-27; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Physical Fitness in Older Adults; Exercise Program
Keywords: physical activity promotion; exercise; physical fitness; elderly; residential care facility
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based exericse program (Experimental): Video-based exercise program "Bliib fit - mach mit!"
  Interventions: Other: Video-based exercise program
- Caregiver-led activation program (Active Comparator): An activation (exercise) program that is instructed and carried out by care professionals as optimized standard care.
  Interventions: Other: Caregiver-led activation program

INTERVENTIONS:
Other: Video-based exercise program — The video-based exercise program - "Bliib fit -mach mit!" focuses on mobilization, muscle strengthening (focus on lower and upper extremities), coordination, balance, and relaxation. Each participant requires the use of a chair for support and to perform exercises in a seated position, if required. The group sessions are supervised by a care professional or registered activation specialist of the residential care facility.
  Arms: Video-based exericse program
Other: Caregiver-led activation program — The caregiver-led activation program (DESKK- Demenzspezifisches Kurzzeitpflegekonzept) is instructed and carried out by care professionals (e.g., nursing staff) as optimized standard care conducted individually or in groups.
  Arms: Caregiver-led activation program

SUMMARY:
The goal of this clinical trial is to learn, if the video-based exercise program "Bliib fit - mach mit!" can be used to improve physical fitness in older adults living in residential care facilities. The main questions it aims to answer are:

Does the video-based exercise program improve participants' physical fitness? Does the video-based exercise program improve participants' quality of life, perceived fall risk, self-efficacy and daily physical activity levels?

Researchers will compare this exercise program to an optimized standard care activation program (caregiver-led) to see if the video-based program can affect physical fitness in older adults living in residential care facilities.

Participants will participate in the exercise or activation program for 12 weeks, four times a week, with each session lasting 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Low to moderate risk of falling
* Physically and cognitively able to independently carry out exercise instructions (based on referral of clinical staff on site)
* Mini Mental State Examination (MMSE) test score ≥ 20

Exclusion Criteria:

* Inability to speak or understand German
* High risk of falling
* Unstable cardiovascular condition or other health condition, which does not support a safe participation in exercise program (based on referral of clinical staff on site, patient file)
* Scheduled transfer to another institution within the next 3 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline, end of intervention at 12 weeks, long-term follow-up 12 weeks after intervention ends
  Lower extremity function and mobility is assessed using the Short Physical Performance Battery (SPPB) (standing balance, gait speed, lower extremity strength). The SPPB is an objective and valid measurement instrument to assess lower extremity function and mobility (> 65 years of age). The measurement instrument consists of three physical tasks: walking, chair-rise-test (sit-to-stand) and standing balance.
Grip strength | Baseline, end of intervention at 12 weeks, long-term follow-up 12 weeks after intervention ends
  Upper extremity strength is assessed using the grip strength test (hand dynamometer). It is a relevant and valid assessment in older adults to assess muscle strength and overall physical function. Participants squeeze a hand dynamometer as hard as they can, three times with each hand.
2-Minutes Walking Test | Baseline, end of intervention at 12 weeks, long-term follow-up 12 weeks after intervention ends
  Aerobic endurance is assessed via the 2-Minutes Walking test. The 2MWT is a submaximal exercise test to assess overall physical fitness and endurance in research and clinical practice. The distance covered in two minutes is recorded. Reference values for adults are available to determine presence of impairments in walking ability, functional endurance, and overall functional status. Oxygen saturation (SpO2) and heart rate (HR) are measured before and after the test using a pulse oximeter. Furthermore, dyspnea and the effort in both legs are measured before and after the test using the Borg scale.

SECONDARY OUTCOMES:
Health-related quality of life | Baseline, end of intervention at 12 weeks, long-term follow-up 12 weeks after intervention ends
  The EuroQol 5-Dimension 5-level (EQ-5D-5L) is a validated 20-item questionnaire to determine health-related quality of life and comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Falls Efficacy Scale | Baseline, end of intervention at 12 weeks, long-term follow-up 12 weeks after intervention ends
  The FES-I Scale is a 16-item questionnaire to measure the concern of falling among older people and addresses various demanding activities inside and outside the home as well as social activities. The levels of concern about falling when carrying out different activities is rated on a four-point scale ranging from 1 = not all concerned to 4= very concerned.
Self-Efficacy | Baseline, end of intervention at 12 weeks, long-term follow-up 12 weeks after intervention ends
  The Exercise Self-Efficacy Scale (ESES) evaluates individuals' confidence in their ability to participate in physical activity and serves as a valuable tool for measuring self-efficacy in this domain. The scale includes six variables and uses a 10-point response scale ranging from "not at all confident" to "very confident," with an option for no response.
Accelerometery | Baseline, end of intervention at 12 weeks, long-term follow-up 12 weeks after intervention ends
  GENEactiv motion sensors (accelerometers) are used to examine daily physical activity levels over seven days. The lightweight device delivers continuous recording of high-resolution acceleration, which enables to classify a person's daily activities in terms of spent lying, sitting, standing, walking (steps), and sleeping. The device places minimal strain on the wearer, is waterproof, and will be worn as a wristband.

CONTACTS AND LOCATIONS:
Overall Officials: Eling de Bruin, Prof., Principal Investigator — Eastern Switzerland University of Applied Sciences
Locations (1):
- Eastern Switzerland University of Applied Sciences, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No